CLINICAL TRIAL: NCT02693873
Title: STOP OA: A PILOT STUDY - Adaptation and Evaluation of a Targeted, Evidence-based, Integrated Patient Education and Exercise Program to Prevent the Progression of Hip and Knee Osteoarthritis Symptoms
Brief Title: STOP OA: A PILOT STUDY (GLA:D Canada) - Education and Targeted, Personalized Exercise for Hip and Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aileen Davis (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other); Arthritis Research Centre of Canada (Other); University of Southern Denmark (Other); Bone and Joint Canada (Unknown)
Responsible Party: Sponsor-Investigator, Aileen Davis, Senior Scientist, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLA:D Canada pilot
Record Dates: First submitted 2016-02-19; First posted 2016-02-29 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis, Hip; Osteoarthritis, Knee; Patient Education; Exercise, Neuromuscular; Disease Management; Evidence-Based Health Care; Pilot Study
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Hip; Osteoarthritis, Knee; Motor Activity | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: GLA:DCanada Program - Education and targeted, personalized exercise for people with hip and/or knee osteoarthritis
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm Study: (Other): All participants will receive GLA:D Canada, an education and neuromuscular exercise program
  Interventions: Behavioral: GLA:D Canada (education and neuromuscular exercise program)

INTERVENTIONS:
Behavioral: GLA:D Canada (education and neuromuscular exercise program) — EDUCATION: 2 sessions cover OA topics (e.g. diagnosis, causes, risk factors, symptoms, treatment). Education also aims to strengthen beliefs in the value of exercise to control and improve pain and encourage exercise adherence after the program.
  EXERCISE: 12 sessions (twice weekly, each about 1-hour) are supervised by therapist(s) with individual progression of exercises when good neuromuscular functioning is demonstrated. Exercises are performed using both legs and focus on sensorimotor control, functional stability, and muscular strength. Exercises involve a 10-minute cycle warm-up followed by a 4-station circuit (i.e. 2 exercises per station with 3 progressive levels of difficulty performed in 2 to 3 sets with 10 to 15 repetitions).
  Other Names: GLA:D (Danish program translated for use in Canada)

SUMMARY:
Osteoarthritis (OA) most often affects the hip and knee joints. The first signs and symptoms of pain, stiffness or swelling are not uncommon in those in their thirties and forties and 10 per cent report symptomatic knee OA by age 60 years. Education and exercise are essential for people with OA to help them manage their condition better. Exercise can reduce pain, improve mobility and enhance quality of life. However, doing the right exercises in the right way is important so that joints are not overly stressed.

The purpose of this study is to evaluate an existing evidence-based program called, Good Life with osteoArthritis in Denmark (GLA:D). The program has been translated and adapted to the Canadian context and will now be implemented in a Canadian therapy setting to start to understand if it is effective. This is the first time this program is being tested in Canada.

While some people have access to self-management programs for OA, these programs often provide only general exercise guidance and education. GLA:D integrates patient education and targeted, personalized exercise for people with hip and/or knee OA. Importantly, the exercises are taught so that individuals learn to incorporate them in their everyday activities. This research is the first step to understanding if people participating in this program have pain relief and improved function and if they are better able to manage their hip or knee OA symptoms. Additionally, this initial evaluation of the program will help create a better understanding of the challenges in delivering the program. This will be valuable information for offering future programs assuming success of this pilot study.

It is anticipated that about 60 people (30 hip OA and 30 knee OA) will participate in this study. These people will be recruited from the Sunnybrook Holland Orthopaedic and Arthritic Centre in Toronto, Ontario, Canada. All consenting participants will receive the GLA:D Canada program delivered by Sunnybrook's therapists.

DETAILED DESCRIPTION:
Arthritis affects over 4.7 million Canadians and the majority of them have hip and/or knee osteoarthritis (OA). Analysis by the Arthritis Alliance of Canada estimates one new OA diagnosis every 60 seconds. Poorly managed OA results in significant pain and disability, reduced quality of life (QOL), limits work productivity and increases use of health care resources. Two of 3 people are under 65 years and 10 percent of people report pain and functional problems from knee OA by age 60 years. Current evidence indicates that education related to OA integrated with exercises targeted to the hip and/or knee joints are effective in reducing symptoms and improving patient function and QOL. Unfortunately, in Canada, while there are some programs for people with bone and joint problems (e.g. OSTEOFIT, Fit & Strong) they are general education and exercise programs and are restricted to people over 60 years. In fact, a recent Bone and Joint Canada workshop identified implementation of evidence-based programs as the number one priority. Additionally, our research showed that people under 60 years are looking for strategies to relieve and prevent OA symptom progression. An evidence-based targeted program integrating patient education and exercise for people with hip and knee OA, Good Life with osteoArthritis in Denmark (GLA:D), was implemented in Denmark by collaborator Roos in 2012. GLA:D is delivered by trained physiotherapists and includes patient education sessions and group exercise twice weekly for six weeks. Importantly, exercises are performed in positions and conditions reflecting daily life emphasizing the quality of performance, proper body position and individualized progression based on the patient's ability. The practical nature of these exercises improves adherence to the exercises in the longer term as they are easily transferrable to daily activities. Feasibility, safety and benefit of GLA:D have been demonstrated in individuals with mild to severe hip and knee OA. Since 2012, more than 5000 patients have been educated in GLA:D. Ongoing benefits for more than 2000 patients with one-year follow-up include pain relief with reduced use of medication, improved function and QOL, return to work, and ongoing use of the new knowledge and skills. Given its successful implementation and outcomes, pilot testing of GLA:D Canada and then potential provincial and national implementation and evaluation is highly appealing to address an urgent need for Canadians with hip and knee OA.

ELIGIBILITY:
Inclusion Criteria:

* 30 years and older
* Hip or knee osteoarthritis diagnosed by a health care provider
* Not a candidate for total joint replacement surgery at the present time
* Fluent in English

Exclusion Criteria:

* Arthritis other than osteoarthritis
* Prior or booked total joint replacement
* Acute knee injury in last 6-months
* Inability to follow instructions and/or to provide consent
* Health condition precluding exercise

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2016-03-07 (Actual); Primary Completion 2016-11-28 (Actual); Study Completion 2017-11-14 (Actual)

PRIMARY OUTCOMES:
Change in hip or knee pain intensity with the Numeric Pain Rating Scale (NPRS) (0 no pain to 10 worst pain imaginable) | Approximately 1-month prior to receiving program (pre-program), 3-months from pre-program, and 12-months from pre-program
  Patient-reported outcome

SECONDARY OUTCOMES:
Arthritis Self-Efficacy Scale (ASES) | Approximately 1-month prior to receiving program (pre-program), 3-months from pre-program, and 12-months from pre-program
  Patient-reported outcome
Hip Disability and Osteoarthritis Outcome Score (HOOS) or the Knee Injury and Osteoarthritis Outcome Score (KOOS) | Approximately 1-month prior to receiving program (pre-program), 3-months from pre-program, and 12-months from pre-program
  Patient-reported outcome
EuroQol - EQ-5D-5L | Approximately 1-month prior to receiving program (pre-program), 3-months from pre-program, and 12-months from pre-program
  Patient-reported outcome
Perceived program benefit | 3-months from pre-program and 12-months from pre-program
  Patient-reported; a single question with five response options ranging from 'not at all beneficial to very beneficial'
Overall program satisfaction | 3-months from pre-program and 12-months from pre-program
  Patient-reported; a single question with five response options ranging from 'not at all satisfied to very satisfied'

OTHER OUTCOMES:
Rapid Assessment of Physical Activity (RAPA) questionnaire | Approximately 1-month prior to receiving program (pre-program), 3-months from pre-program, and 12-months from pre-program
  Patient-reported outcome
Patient Knowledge Questionnaire - Osteoarthritis (PKQ-OA) | Approximately 1-month prior to receiving program (pre-program), 3-months from pre-program, and 12-months from pre-program
  Patient-reported outcome
Number of days in a typical week with at least 30 minutes of physical activity | Approximately 1-month prior to receiving program (pre-program), 3-months from pre-program, and 12-months from pre-program
  Patient-reported outcome
30-second chair stand test | Baseline and 3-months from pre-program
  Administered by the therapist delivering GLA:D
40-metre walk test | Baseline and 3-months from pre-program
  Administered by the therapist delivering GLA:D

CONTACTS AND LOCATIONS:
Overall Officials: Aileen M Davis, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Holland Orthopaedic & Arthritic Centre, Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available.

REFERENCES:
- [Background] O'Donnell S, Lagace C, McRae L, Bancej C. Life with arthritis in Canada: a personal and public health challenge. Chronic Dis Inj Can. 2011 Jun;31(3):135-6. PMID 21733351
- [Background] McAlindon TE, Bannuru RR, Sullivan MC, Arden NK, Berenbaum F, Bierma-Zeinstra SM, Hawker GA, Henrotin Y, Hunter DJ, Kawaguchi H, Kwoh K, Lohmander S, Rannou F, Roos EM, Underwood M. OARSI guidelines for the non-surgical management of knee osteoarthritis. Osteoarthritis Cartilage. 2014 Mar;22(3):363-88. doi: 10.1016/j.joca.2014.01.003. Epub 2014 Jan 24. PMID 24462672
- [Background] Fernandes L, Hagen KB, Bijlsma JW, Andreassen O, Christensen P, Conaghan PG, Doherty M, Geenen R, Hammond A, Kjeken I, Lohmander LS, Lund H, Mallen CD, Nava T, Oliver S, Pavelka K, Pitsillidou I, da Silva JA, de la Torre J, Zanoli G, Vliet Vlieland TP; European League Against Rheumatism (EULAR). EULAR recommendations for the non-pharmacological core management of hip and knee osteoarthritis. Ann Rheum Dis. 2013 Jul;72(7):1125-35. doi: 10.1136/annrheumdis-2012-202745. Epub 2013 Apr 17. PMID 23595142
- [Background] Dunlop DD, Song J, Semanik PA, Chang RW, Sharma L, Bathon JM, Eaton CB, Hochberg MC, Jackson RD, Kwoh CK, Mysiw WJ, Nevitt MC, Hootman JM. Objective physical activity measurement in the osteoarthritis initiative: Are guidelines being met? Arthritis Rheum. 2011 Nov;63(11):3372-82. doi: 10.1002/art.30562. PMID 21792835
- [Background] Nuesch E, Dieppe P, Reichenbach S, Williams S, Iff S, Juni P. All cause and disease specific mortality in patients with knee or hip osteoarthritis: population based cohort study. BMJ. 2011 Mar 8;342:d1165. doi: 10.1136/bmj.d1165. PMID 21385807
- [Background] Hawker GA, Croxford R, Bierman AS, Harvey PJ, Ravi B, Stanaitis I, Lipscombe LL. All-cause mortality and serious cardiovascular events in people with hip and knee osteoarthritis: a population based cohort study. PLoS One. 2014 Mar 7;9(3):e91286. doi: 10.1371/journal.pone.0091286. eCollection 2014. PMID 24608134
- [Background] Rissanen P, Aro S, Sintonen H, Asikainen K, Slatis P, Paavolainen P. Costs and cost-effectiveness in hip and knee replacements. A prospective study. Int J Technol Assess Health Care. 1997 Fall;13(4):575-88. doi: 10.1017/s0266462300010059. PMID 9489250
- [Background] Gunther KP. Surgical approaches for osteoarthritis. Best Pract Res Clin Rheumatol. 2001 Oct;15(4):627-43. doi: 10.1053/berh.2001.0178. PMID 11567544
- [Background] Felts W, Yelin E. The economic impact of the rheumatic diseases in the United States. J Rheumatol. 1989 Jul;16(7):867-84. PMID 2527991
- [Background] Centers for Disease Control and Prevention (CDC). Prevalence of doctor-diagnosed arthritis and arthritis-attributable activity limitation--United States, 2010-2012. MMWR Morb Mortal Wkly Rep. 2013 Nov 8;62(44):869-73. PMID 24196662
- [Background] Losina E, Weinstein AM, Reichmann WM, Burbine SA, Solomon DH, Daigle ME, Rome BN, Chen SP, Hunter DJ, Suter LG, Jordan JM, Katz JN. Lifetime risk and age at diagnosis of symptomatic knee osteoarthritis in the US. Arthritis Care Res (Hoboken). 2013 May;65(5):703-11. doi: 10.1002/acr.21898. PMID 23203864
- [Background] Bennell KL, Hunt MA, Wrigley TV, Lim BW, Hinman RS. Role of muscle in the genesis and management of knee osteoarthritis. Rheum Dis Clin North Am. 2008 Aug;34(3):731-54. doi: 10.1016/j.rdc.2008.05.005. PMID 18687280
- [Background] Brandt KD, Dieppe P, Radin EL. Etiopathogenesis of osteoarthritis. Rheum Dis Clin North Am. 2008 Aug;34(3):531-59. doi: 10.1016/j.rdc.2008.05.011. PMID 18687271
- [Background] Rutherford DJ, Hubley-Kozey CL, Stanish WD. Changes in knee joint muscle activation patterns during walking associated with increased structural severity in knee osteoarthritis. J Electromyogr Kinesiol. 2013 Jun;23(3):704-11. doi: 10.1016/j.jelekin.2013.01.003. Epub 2013 Jan 26. PMID 23357547
- [Background] Fitzgerald GK, Piva SR, Irrgang JJ. Reports of joint instability in knee osteoarthritis: its prevalence and relationship to physical function. Arthritis Rheum. 2004 Dec 15;51(6):941-6. doi: 10.1002/art.20825. PMID 15593258
- [Background] Ageberg E. Consequences of a ligament injury on neuromuscular function and relevance to rehabilitation - using the anterior cruciate ligament-injured knee as model. J Electromyogr Kinesiol. 2002 Jun;12(3):205-12. doi: 10.1016/s1050-6411(02)00022-6. PMID 12086815
- [Background] Skou ST, Simonsen ME, Odgaard A, Roos EM. Predictors of long-term effect from education and exercise in patients with knee and hip pain. Dan Med J. 2014 Jul;61(7):A4867. PMID 25123117
- [Background] Skou ST, Odgaard A, Rasmussen JO, Roos EM. Group education and exercise is feasible in knee and hip osteoarthritis. Dan Med J. 2012 Dec;59(12):A4554. PMID 23290290
- [Background] Ageberg E, Link A, Roos EM. Feasibility of neuromuscular training in patients with severe hip or knee OA: the individualized goal-based NEMEX-TJR training program. BMC Musculoskelet Disord. 2010 Jun 17;11:126. doi: 10.1186/1471-2474-11-126. PMID 20565735
- [Background] Hill J, Bird H. Patient knowledge and misconceptions of osteoarthritis assessed by a validated self-completed knowledge questionnaire (PKQ-OA). Rheumatology (Oxford). 2007 May;46(5):796-800. doi: 10.1093/rheumatology/kel407. Epub 2006 Dec 18. PMID 17178737
- [Background] Jensen MP, McFarland CA. Increasing the reliability and validity of pain intensity measurement in chronic pain patients. Pain. 1993 Nov;55(2):195-203. doi: 10.1016/0304-3959(93)90148-I. PMID 8309709
- [Background] Williamson A, Hoggart B. Pain: a review of three commonly used pain rating scales. J Clin Nurs. 2005 Aug;14(7):798-804. doi: 10.1111/j.1365-2702.2005.01121.x. PMID 16000093
- [Background] Lorig K, Chastain RL, Ung E, Shoor S, Holman HR. Development and evaluation of a scale to measure perceived self-efficacy in people with arthritis. Arthritis Rheum. 1989 Jan;32(1):37-44. doi: 10.1002/anr.1780320107. PMID 2912463
- [Background] Lorig K, Holman H. Arthritis Self-Efficacy Scales measure self-efficacy. Arthritis Care Res. 1998 Jun;11(3):155-7. doi: 10.1002/art.1790110302. No abstract available. PMID 9782806
- [Background] Topolski TD, LoGerfo J, Patrick DL, Williams B, Walwick J, Patrick MB. The Rapid Assessment of Physical Activity (RAPA) among older adults. Prev Chronic Dis. 2006 Oct;3(4):A118. Epub 2006 Sep 15. PMID 16978493
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Bredin SS, Gledhill N, Jamnik VK, Warburton DE. PAR-Q+ and ePARmed-X+: new risk stratification and physical activity clearance strategy for physicians and patients alike. Can Fam Physician. 2013 Mar;59(3):273-7. No abstract available. PMID 23486800
- See also: Click here for more information about the GLA:D program. Working with researchers from Denmark, Bone and Joint Canada has launched the "GLA:D Canada" program at Sunnybrook Health Sciences Centre. — http://boneandjointcanada.com/osteoarthritis/health-care-professionals/glad-canada/